CLINICAL TRIAL: NCT03875170
Title: Efficacy of an Intervention by Proprioceptive Neuromuscular Facilitation in the Flexibility and Strength of Flexor Muscles and Hamstrings, in Federated Football Players From 18 to 30 Years Old. A Randomized Clinical Trial.
Brief Title: Proprioceptive Neuromuscular Facilitation in the Flexibility and Strength of Flexor Muscles and Hamstrings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FNP
Record Dates: First submitted 2019-03-10; First posted 2019-03-14 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Proprioceptive Disorders
Keywords: Proprioceptive Neuromuscular Facilitation; Range of motion; Stretching; Muscle strength; Randomized clinical trial
MeSH Terms: conditions — Somatosensory Disorders | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive neuromuscular facilitation (Experimental): Each session will last 5 minutes for each subject, taking place two sessions a week, in a period of 6 weeks. The intervention will be made at the beginning of the training session. The technique will be carried out with the subjects in the positions of supine, prone and lateral position, for the flexor muscles of the hip, hamstrings and quadriceps, where the musculature and the joint to be treated will be taken to a range of functional mobility
  Interventions: Other: Experimental
- Muscle stretching (Active Comparator): Each session will last 5 minutes for each subject, taking place two sessions a week, in a period of 6 weeks. The intervention will be made at the beginning of the training session. It will be done for the hip, quadriceps and hamstring muscles with a voluntary antagonist activation to relax the agonist muscle.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The technique will be carried out with the subjects in the positions of supine, prone and lateral position, for the flexor muscles of the hip, hamstrings and quadriceps, where the musculature and the joint to be treated will be taken to a range of functional mobility. The subject will be asked to perform an isometric contraction, with a series of 3 seconds for sustained contraction and a rest between contraction of 2 to 3 seconds after activating the Golgi apparatus, making an inhibition of the stimulus and bringing the joint and muscle to the highest possible range of motion without pain.
  Other Names: Proprioceptive neuromuscular facilitation
  Arms: Proprioceptive neuromuscular facilitation
Other: Control — The active stretching technique will be performed for the hip, quadriceps and hamstring flexors with a voluntary antagonist activation to relax the agonist muscle, holding the movement to be performed for 30 seconds to stimulate the neuromuscular spindle and produce a relaxation of the muscle fibers.
  Other Names: Muscle stretching
  Arms: Muscle stretching

SUMMARY:
Introduction: The loss of normal values of ROM due to the lack of flexibility and strength in the hip flexors, quadriceps and hamstrings in soccer players can cause a loss of mobility of the hip and knee joint. Proprioceptive neuromuscular facilitation is an active-assisted stretching technique used to improve flexibility and therefore the ranges of joint mobility.

Aim. To assess the effectiveness of an intervention by proprioceptive neuromuscular facilitation in the improvement of flexibility and strength in the hamstring, hip flexor and quadriceps musculature compared to conventional stretches in football players.

Study design. Randomized, multicentric, single-blind clinical study. Methods. The 30 players will be randomly assigned to the study groups: experimental (proprioceptive neuromuscular facilitation and static stretches) and control (static stretches). The treatment will last 6 weeks, with two sessions a week of 5 minutes each. The study variables will be the range of hip mobility (using goniometry), hamstring flexibility (using the EPR test, inclinometer) and the strength of hip flexors, quadriceps and hamstrings (through the RM test). A descriptive statistical analysis will be carried out calculating the main statistical characteristics and after calculating the normality of the sample (test Kolmogorov- Smirnov), the differences between evaluations in each group (t-student test) and the intra- and intersubject effect will be calculated (ANOVA of repeated measures).

Expected results. Improved hip mobility, hamstring flexibility and strength in hip flexors, quadriceps and hamstrings muscles.

ELIGIBILITY:
Inclusion Criteria:

* Volleyball players
* Male
* From 18 to 30 years old
* Federated in the Royal Federation of Football of the Community of Madrid
* Not had any musculoskeletal injuries in the last 3 months.

Exclusion Criteria:

* Impossibility, for work or academic reasons, to comply with the requirements of the study (interventions and evaluations);
* Under pharmacological treatment
* Who are exercising a physiotherapy treatment parallel to the development of the study
* Not sign the informed consent document.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline flexibility of the hamstring muscles after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The measurement instrument to measure the flexibility of the hamstring muscles is the passive elevation of the straight leg with an inclinometer (model ISOMED, Inc., Portland, OR) to be placed on the tibia (as distal as possible). The physiotherapist will maintain the extension of the knee and the leg will be lifted by the evaluator to a hip flexion, until the subject indicates pain in the hamstring muscles, when the evaluator perceives hip flexion restriction or when a posterior pelvic tilt occurs. The contralateral knee of the subject will remain in extension. The unit of measurement of the test is the maximum angle read from the inclinometer at the point of maximum flexibility, in degrees, with the normative range of 75 to 80 degrees (the greater the degree of flexibility, the greater the flexibility).

SECONDARY OUTCOMES:
Change from baseline the range of motion of hip after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The range of motion of the hip will be evaluated using a universal long arm goniometer. The hip flexion will be measured with the goniometer as the deviation from the neutral zero position in which the lower extremity and the trunk are in the horizontal plane. The fixed arm of the goniometer will be aligned on the horizontal axis of the body, while the mobile arm of the goniometer will be aligned on the lateral midline of the thigh, placing the goniometer support axis on the greater trochanter. Hip adduction and hip abduction will be measured from the neutral zero position in which the longitudinal axis of the thigh is perpendicular to the transverse line through the anterior superior iliac spines of the pelvis. The contralateral leg will be hanging over the edge of the stretcher. The unit of measurement for this test is the grade, with a range of normative movement from 0 to 50 degrees (the higher the graduation, the greater the mobility of the hip).
Change from baseline strength of upper limbs after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The strength of upper limbs will be measured with the 1RM test. This test is defined as the maximum repetition with the heaviest load through a full range of motion. To calculate the 1 RM, the indirect relationship methods of lifting a submaximal load with a full range of motion to failure will be used. From this action a mathematical model related to the load and the number of repetitions until the failure will be made, obtaining a value of force. The unit of measurement of this evaluation is the kilogram (a higher value indicates a greater performance in the strength of lower limbs)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- European University of Madrid, Madrid, Spain